CLINICAL TRIAL: NCT04715633
Title: PD-1 Inhibitors (Camrelizumab) Combined With VEGF Inhibitors (Apatinib) for Locally Advanced dMMR/MSI-H Colorectal Cancer: an Open-label, Multi-center, Phase II Clinical Trial
Brief Title: PD-1 Inhibitors Combined With VEGF Inhibitors for Locally Advanced dMMR/MSI-H Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangdong Provincial People's Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Pei-Rong Ding, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-120-03
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer; Microsatellite Instability High
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Immune Checkpoint Inhibitors; camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 inhibitors plus VEGF inhibitors (Experimental): Patients will be given 4 cycles of Camrelizumab (200mg iv every 3 weeks) plus Apatinib (250mg QD day1-14) before being evaluated for response.
  Interventions: Drug: PD-1 inhibitor plus VEGF inhibitors

INTERVENTIONS:
Drug: PD-1 inhibitor plus VEGF inhibitors — Camrelizumab 200mg IV every 3 weeks; Apatinib 250mg QD day 1-14. Rescue chemotherapy: Oxaliplatin 130mg/m2 IV drip Q3W d1+Capecitabine 1000mg/m2 QD d1-d14 Rescue chemoradiotherapy: Long-course radiotherapy +Capecitabine 825mg/m2 QD d1-d14
  Other Names: Camrelizumab plus Apatinib

SUMMARY:
In this open-label phase II study, patients will be scheduled for neoadjuvant treatment with PD-1 inhibitors (Camrelizumab) plus VEGF inhibitor (Apatinib) for dMMR/MSI-H colorectal cancer staged as locally advanced (cT3-4N+/-M0 for rectal cancer, cT4 or cT3 with extramural extension ≥5mm for colon cancer). Radiological evaluation will be preformed after 4 cycles of treatment. Patients (either with colon or rectal cancer) who achieve complete clinical response will be offered the choice of Watch & Wait.

DETAILED DESCRIPTION:
This is an open-label phase II study, with the aim of determining the efficacy of PD-1 inhibitors (Camrelizumab) plus VEGF inhibitor (Apatinib) as a neoadjuvant therapy for dMMR/MSI-H locally advanced colorectal cancer.

Patients will be evaluated for eligibility within 14 days prior to study initiation with CT (for colon cancer) and/or MRI (for rectal cancer).

Patients will be given four cycles of Camrelizumab (200mg iv every 3 weeks) plus Apatinib (250mg QD day1-14) before being evaluated for response. For patients with colon cancer, if a SD/PD is achieved and the tumor is deemed unresectable, they will be offered chemotherapy±radiotherapy, while if a CR or PR is achieved, they will be offered another four cycles of Camrelizumab + Apatinib. After completing 8 cycles of treatment, if a CR is achieved they will be offered the choice of Watch & Wait. For patients with rectal cancer who have a SD/PD (after 4 cycles), chemoradiotherapy will be offered, while for those with a CR/PR, another four cycles of the treatment will be given. After completing 8 cycles of treatment, if a CR is achieved patients will be offered the choice of Watch & Wait.

ELIGIBILITY:
Inclusion Criteria:

* Locally confirmed dMMR or MSI-H colorectal carcinoma
* Tumor staging based on CT/MR or transrectal ultrasound imaging:
* Colon cancer: radiological high risk (rT4 or rT3 tumour with extramural extension ≥ 5mm with or without lymph node involvement)
* Rectal cancer: <12 cm from the anal verge and radiological high risk (rT3/4 with or without lymph node involvement)
* No sign of bowel obstruction, or bowel obstruction has been relieved by ostomy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 10 days prior to study start
* Aged 18 or over
* Life expectancy of at least 2 years
* Measurable disease
* Female participants of childbearing potential must be willing to use adequate contraception for the course of the study starting with the first dose of study medication through 120 days after the last PD-1 antibody dose
* Male participants must agree to use adequate contraception for the course of the study starting with the first dose of study medication through 120 days after the last PD-1 antibody dose
* Adequate organ function

Exclusion Criteria:

* Active autoimmune disease that has required systemic treatment in past 2 years
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 2 weeks prior to this study start
* Currently participating and receiving treatment in another study within 4 weeks of study start
* History of severe allergic reaction to monoclonal antibody
* Strong evidence of distant metastases or peritoneal nodules (M1)
* Colonic obstruction that has not been defunctioned
* Has received prior therapy with an immune checkpoint inhibitor (e.g., anti-programmed cell death [PD]-1, anti-PD ligand 1 [L1], anti-PD-L2 agent, or anti-cytotoxic T-lymphocyte-associated protein 4 [CTLA-4] agent, etc.) or anti-VEGF agents (e.g., Bevacizumab, Apatinib)
* Any other malignant disease within the preceding 5 years with the exception of non-melanomatous skin cancer, carcinoma in situ and early stage disease with a recurrence risk <5%
* Received a live vaccine within 30 days of planned start of study medication
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis B or C
* Known history of, or any evidence of interstitial lung disease or active, non-infectious pneumonitis
* Known history of active tuberculosis (Bacillus tuberculosis [TB])
* Active infection requiring systemic therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response or pathological complete response | up to 2 year
  Clinical complete response or immunotherapy-related pathological complete response (cCR or immunotherapy-related pCR)

SECONDARY OUTCOMES:
Objective Response Rate (ORR, PR+CR) | up to 2 year
  Partial response + complete response
3-year relapse-free survival | up to 3 years
3-year overall survival | up to 3 years
Surgical complications | within 1 month after surgery
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Rong Ding, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- 651 Dongfeng Road East, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yu JH, Xiao BY, Li DD, Jiang W, Ding Y, Wu XJ, Zhang RX, Lin JZ, Wang W, Han K, Kong LH, Zhang XK, Chen BY, Mei WJ, Pan ZZ, Tang JH, Zhang XS, Ding PR. Neoadjuvant camrelizumab plus apatinib for locally advanced microsatellite instability-high or mismatch repair-deficient colorectal cancer (NEOCAP): a single-arm, open-label, phase 2 study. Lancet Oncol. 2024 Jul;25(7):843-852. doi: 10.1016/S1470-2045(24)00203-1. Epub 2024 Jun 6. PMID 38852601